CLINICAL TRIAL: NCT03173170
Title: A Single-Sequence, Open-Label, 2-Period Crossover Trial to Evaluate the Effect of the Potent Cytochrome P-450 3A4 Inhibitor Itraconazole on the Pharmacokinetics of TAK-954 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of the Potent Cytochrome P-450 3A4 (CYP3A4) Inhibitor Itraconazole on the Pharmacokinetics (PK) of TAK-954 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-954-1004; 2017-000713-22 (EudraCT Number); U1111-1195-7682 (Registry Identifier: WHO)
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants
Keywords: Drug Therapy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg (Experimental): TAK-954 0.2 milligram (mg), infusion, intravenously, once on Day 1 of First Intervention Period, followed by a minimum of 7-day washout period, further followed by Itraconazole 200 mg, capsule, orally, once daily on Days 1 to 8 along with TAK-954 0.2 mg, infusion, intravenously on Day 4 of Second Intervention Period.
  Interventions: Drug: TAK-954; Drug: Itraconazole

INTERVENTIONS:
Drug: TAK-954 — TAK-954 Infusion
Drug: Itraconazole — Itraconazole Capsule

SUMMARY:
The purpose of this study is to evaluate the effect of the potent CYP3A4 inhibitor itraconazole on the single-dose PK of TAK-954.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. TAK-954 is being tested in healthy participants in order to evaluate the effect of the potent CYP3A4 inhibitor itraconazole on the single-dose PK of TAK-954.

The study will enroll approximately 10 participants. Participants will receive the following treatment sequences:

• TAK-954 0.2 mg; Itraconazole 200 mg + TAK-954 0.2 mg

Participants will be given an intravenous infusion of TAK-954 on Day 1 of First Intervention Period (6 days) followed by minimum 7-day washout period, after which participants will be given Itraconazole capsule on Days 1 to 8 along with TAK-945 infusion on Day 4 of Second Intervention Period (9 days).

This single center trial will be conducted in the United States. The overall duration to participate in this study is 7 to 8 weeks. Participants will visit the clinic on Day -1 and remained confined until Day 6 (First Intervention Period) and Day 9 (Second Intervention Period). Participants will return for a Follow-up Visit 10 to 14 days after last dose of study drug (approximately up to Day 34).

ELIGIBILITY:
Inclusion Criteria:

1. Is a man or woman (with no child bearing potential) aged 18 to 55 years, inclusive, at the Screening Visit.
2. Has a body mass index (BMI) from greater than or equal to (>=) 18 and less than or equal to (<=) 30 kilogram per square meter (kg/m^2) and has a body weight greater than (>) 50 kilogram (kg) at the Screening Visit.
3. Is a nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before administration of the initial dose of trial drug/invasive procedure.

Exclusion Criteria:

1. Has a positive alcohol or drug screen.
2. Had major surgery, donated or lost 1 unit of blood (approximately 500 milliliter (mL)) within 8 weeks of the first dose of study drug.
3. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).
4. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
5. Has a substance abuse disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Pharmaceutical Research Associates, Inc., Lenexa, Kansas, United States

REFERENCES:
- [Derived] Chen C, Zhang L, Almansa C, Rosario M, Cwik M, Balani SK, Lock R. Evaluation of the Pharmacokinetics of Felcisetrag (TAK-954), a 5-HT4 Receptor Agonist, in the Presence and Absence of Itraconazole, a Potent CYP3A4 Inhibitor. Clin Pharmacol Drug Dev. 2022 Feb;11(2):142-149. doi: 10.1002/cpdd.1046. Epub 2022 Jan 6. PMID 34989180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United States from 31 May 2017 to 24 July 2017.
Pre-assignment Details: Healthy participants were enrolled in this single sequence 2-period crossover study to receive TAK-954 0.2 milligram (mg) in Intervention Period 1 followed by itraconazole 200 mg + TAK-954 0.2 mg in Intervention Period 2.
Groups:
- TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg: TAK-954 0.2 mg, infusion, intravenously, once on Day 1 of First Intervention Period, followed by a minimum of 7-day washout period, further followed by itraconazole 200 mg, capsule, orally, once daily on Days 1 to 8 along with TAK-954 0.2 mg, infusion, intravenously on Day 4 of Second Intervention Period.
Period: First Intervention Period (6 Days)
Arm/Group | TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg
Started | 10
Completed | 10
Not Completed | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg
Started | 10
Completed | 10
Not Completed | 0
Period: Intervention Period 2 (9 Days)
Arm/Group | TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | TAK-954 0.2 mg + Itraconazole 200 mg and TAK-954 0.2mg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.72 (11.534)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 174.4 (10.17)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.2 (2.90)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-954
Time Frame: TAK-954 0.2 mg: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose; Itraconazole 200 mg and TAK-954 0.2 mg: Day 4 pre-dose and at multiple time points (up to 120 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- TAK-954 0.2 mg: TAK-954 0.2 mg, infusion, intravenously, once on Day 1 of First Intervention Period.
- Itraconazole 200 mg and TAK-954 0.2 mg: Itraconazole 200 mg, capsule, orally, once daily on Days 1 to 8 along with TAK-954 0.2 mg, infusion, intravenously on Day 4 of Second Intervention Period.
Arm/Group | TAK-954 0.2 mg | Itraconazole 200 mg and TAK-954 0.2 mg
Number analyzed (Participants) | 10 | 10
nanogram/milliliter (ng/mL) | 2.642 (0.4426) | 2.840 (0.6497)
Statistical Analysis 1: Comparison: TAK-954 0.2 mg vs Itraconazole 200 mg and TAK-954 0.2 mg; A paired t-test on the natural log-transformed parameters was performed. The means and difference of means for the log-transformed parameters were exponentiated to obtain the point estimates of the itraconazole effect and 90 percent (%) confidence intervals (CIs); Test type: Other; Mean ratio = 1.0622, 90% CI 2-sided [0.9569 to 1.1792]

2. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-954
Time Frame: TAK-954 0.2 mg: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose; Itraconazole 200 mg and TAK-954 0.2mg: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose
Population: The PK set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration. PK analysis set where Day 1 and 4 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Groups:
- Itraconazole 200 mg and TAK-954 0.2mg: Itraconazole 200 mg, capsule, orally, once daily on Days 1 to 8 along with TAK-954 0.2 mg, infusion, intravenously on Day 4 of Second Intervention Period.
Arm/Group | TAK-954 0.2 mg | Itraconazole 200 mg and TAK-954 0.2mg
Number analyzed (Participants) | 10 | 10
hour*nanogram per milliliter (hr*ng/mL) | 28.59 (6.550) | 43.15 (10.265)
Statistical Analysis 1: Comparison: TAK-954 0.2 mg vs Itraconazole 200 mg and TAK-954 0.2mg; A paired t-test on the natural log-transformed parameters was performed. The means and difference of means for the log-transformed parameters were exponentiated to obtain the point estimates of the itraconazole effect and 90% CIs; Test type: Other; Mean ratio = 1.4892, 90% CI 2-sided [1.3851 to 1.6012]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to Day 9 of Second Intervention Period
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Itraconazole 200 mg: Itraconazole 200 mg, capsule, orally, once daily on Days 1 to 3 of Second Intervention Period.
- Itraconazole 200 mg and TAK-954 0.2 mg: Itraconazole 200 mg, capsule, orally, once daily on Days 4 to 8 along with TAK-954 0.2 mg, infusion, intravenously on Day 4 of Second Intervention Period.
Arm/Group | TAK-954 0.2 mg | Itraconazole 200 mg | Itraconazole 200 mg and TAK-954 0.2 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-954 0.2 mg (N=10) | Itraconazole 200 mg (N=10) | Itraconazole 200 mg and TAK-954 0.2 mg (N=10)
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03173170/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT03173170/SAP_001.pdf